CLINICAL TRIAL: NCT03914001
Title: Comprehensive Multiparametric Magnetic Resonance Imaging After Transurethral Resection of Non Muscle-invasive Bladder Tumor; Can it Replace Second Look Biopsy? A Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE 2390
Record Dates: First submitted 2019-04-06; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Bladder Cancer
Keywords: Non muscle invasive bladder cancer; multiparametric magnetic resonance imaging; second resection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMIBC patients (Other): eligible patients will undergo initial mpMRI before initial TURBT, then followed by second mpMRI and second resection TURBT after 4 weeks
  Interventions: Device: mpMRI; Procedure: Second look TURBT

INTERVENTIONS:
Device: mpMRI — all eligible patients will undergo mpMRI 4 weks after initial TURBT
Procedure: Second look TURBT — after mpMRI all patients will subjected to second look TURBT

SUMMARY:
The aim of the study is to prospectively assess the role of mpMRI as a non invasive method for assessment of possible residual tumor after initial resection of non muscle invasive bladder tumor.

DETAILED DESCRIPTION:
Comprehensive multiparametric (mp) MRI which includes T2 weighted imaging, dynamic contrast enhanced (DCE) imaging and DWI, was proven to be efficient tool in differentiating benign and malignant bladder lesion. morphological characterization of malignant bladder lesion (mapping/size/morphology/stalk), T stage differentiation and histological grade discrimination.

The application of mpMRI in NMIBC with its added value as non invasive tool for initial staging and after primary resection could be a new helpful method for better diagnosis, risk categorization, refining the indications of second resection and proper determination of adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Patients with primary or recurrent papillary NMIBC.
3. Normal cardiac, hematological, and renal functions.

Exclusion Criteria:

* 1. Patients with history of previous radiotherapy or systemic chemotherapy. 2. Patients suffering from immuno-deficiency or other malignancies. 3. Patients with high serum creatinine (more than 2 mg/dl). 4. Patients with contraindication to MRI (claustrophobia-pacemaker- metallic prosthesis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
assessment of the performance of mpMRI as a diagnostic tool for possible residual malignancy after initial TURBT | 1 year
  assessment of the performance of mpMRI as a diagnostic tool for possible residual malignancy after initial TURBT by comparing the results obtained by pre-second look TURBT mpMRI (Test of the study) with results of second look biopsy whether benign or malignant (Standard test).

SECONDARY OUTCOMES:
Predictive capability of initial mpMRI of differentiation between benign and malignant bladder lesions. | 1 year
  Predictive capability of initial mpMRI of differentiation between benign and malignant bladder lesions.
2- Predictive capability of initial mpMRI of differentiation between NMIBC and muscle invasive disease. | 1 year
  2- Predictive capability of initial mpMRI of differentiation between NMIBC and muscle invasive disease.
Accuracy of bladder mapping in initial mpMRI (18) as a guide during TURBT. | 1 year
  Accuracy of bladder mapping in initial mpMRI (18) as a guide during TURBT.
Predictive value of initial mpMRI for characterization of NMIBC (T stage, Grading, Risk categorization). | 1 year
  Predictive value of initial mpMRI for characterization of NMIBC (T stage, Grading, Risk categorization).
Rate of over staging and under staging of NMIBC after second look TURBT in this prospective series. | 1 year
  Rate of over staging and under staging of NMIBC after second look TURBT in this prospective series.
Morbidity (using modified Dindo-Clavian system for post-operative complications (19) and mortality rates after second look TURBT. | 1 year
  Morbidity (using modified Dindo-Clavian system for post-operative complications (19) and mortality rates after second look TURBT.
Readmission rate after second look TURBT. | 1 year
  Readmission rate after second look TURBT.
Cost comparison of mpMRI and second look TURBT. | 1 year
  Cost comparison of mpMRI and second look TURBT.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, Study Chair — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt